CLINICAL TRIAL: NCT06266949
Title: Perimetry Based on Eye-movements in Patients With (Supra)Sellar Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11362
Record Dates: First submitted 2024-01-25; First posted 2024-02-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-05

CONDITIONS: Pituitary Tumor; Visual Fields Hemianopsia
MeSH Terms: conditions — Pituitary Neoplasms; Hemianopsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Participants will undergo a visual acuity test. Next they will perform the SONDA test 2 times at one visit and once more in a later visit Participants will fill in a questionnaire
  Interventions: Diagnostic Test: SONDA
- Healthy controls: Participants will perform the SONDA test 2 times
  Interventions: Diagnostic Test: SONDA

INTERVENTIONS:
Diagnostic Test: SONDA — Perimetry based visualfield analysis

SUMMARY:
The purpose of this study is to assess wether the SONDA visual field test is suitable for patients with a supra sellar tumour.

DETAILED DESCRIPTION:
The objective of this study is to determine whether SONDA is non-inferior in predicting visual field limitations compared to the SAP in patients with a (supra)sellar tumor. The study population will be made up of patients with a (supra)sellar tumor complicated by compression of the optic chiasm as well as healthy controls. The patients will be asked to join the study when the patients are referred to the UMCG for further diagnostics and treatment. In case the patients show signs of visual field loss the patients will be asked to participate in the study. The researchers will reuse data from healthy controls collected in previous studies where possible and, if necessary for age matching, recruit new participants. Participants will be asked to perform the SONDA test before and after surgery. The first time the participants will perform the test twice and will also perform routine eye test and be asked to fill in a questionnaire to evaluate the experience.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a (supra)sellar tumor
* Visual field loss based on the most recent SAP; False positive rate <15%; fixation losses <20%
* Informed written consent

Exclusion Criteria:

* Neurological disorders
* Eye disease not related to a (supra)sellar tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a (supra)sellar tumour and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Convert validity | Baseline
  Difference (dB) between the predicted MD (SONDA) and the assessed MD (SAP), expressed as delta MD.
Test-retest reliability | baseline 1, baseline 2, 6-8 weeks post-operative
  The variability of the predicted MD (dB) between consecutive measurements in the same person.

SECONDARY OUTCOMES:
Experience | Baseline
  The experience of patients expressed in scores and descriptives based on a questionnaire: Questionnaire Standardized Oculomotor and Neuro-Ophthalmic Disorder Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jos MA Kuijlen, MD/PHD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided